CLINICAL TRIAL: NCT02880722
Title: Development and Validation of a Real-time Patient-Reported Outcome Measure for Chronic Abdominal Pain: The Experience Sampling Method (ESM)
Brief Title: Experience Sampling Method for Symptom Assessment in Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NL57473.068.16
Record Dates: First submitted 2016-07-28; First posted 2016-08-26 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome (IBS); Experience Sampling Method (ESM); Ecological Momentary Assessment (EMA); Abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IBS patients: IBS according to Rome IV criteria.
- Healthy control group: Healthy volunteers without abdominal complaints fulfilling Rome IV criteria for IBS.

SUMMARY:
Reliable patient reported outcome measures (PROM's) for symptom assessment in irritable bowel syndrome are essential in order to investigate natural disease course and potential treatment options aimed at symptom improvement, since biological markers are currently unavailable. Currently used symptom assessment methods, i.e. end-of-day or end-of-week questionnaires, have considerable limitations. The Experience Sampling Method (ESM), an electronic questioning method characterized by random and repeated, momentary assessments in the subject's current state and environment, might overcome these limitations. Aim of this study is to validate an IBS-specific electronic patient-reported outcome measure, based on the Experience Sampling Method-principle, for symptom assessment in IBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of irritable bowel syndrome according to Rome IV criteria.
* Ability to understand and speak the national language of the concerning center.
* Ability to understand how to utilize the ESM-tool.

Exclusion Criteria:

* Any organic explanation for the abdominal complaints.
* A history of abdominal surgery, except for uncomplicated appendectomy, laparoscopic cholecystectomy and hysterectomy.
* Start up of regularly used medication from one month before inclusion until the end of study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBS patients.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Abdominal pain scores as measured by the ESM tool. | 7 days
  Momentary measurements.

SECONDARY OUTCOMES:
Abdominal pain scores as measured by the end-of-day diary. | 7 days
  Retrospective measurements with a recall period of one day.
Abdominal pain scores as measured by the Gastrointestinal Symptom Rating Scale - IBS. | 7 days
  Retrospective measurements with a recall period of one week.
Symptom scores (other than abdominal pain) as measured using the ESM-tool. | 7 days
  Gastrointestinal symptoms, psychological symptoms, extra-intestinal symptoms, data on context and environment.
Gastrointestinal symptom scores (other than abdominal pain) as measured using the end-of-day diary. | 7 days
Gastrointestinal symptom scores (other than abdominal pain) as measured using the GSRS-IBS. | 7 days
Psychological symptom scores as measured using the PHQ-9. | 7 days
Psychological symptom scores as measured using the GAD-7. | 7 days
Quality of life scores as measured using SF-36. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ad A.M. Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided